CLINICAL TRIAL: NCT05860751
Title: The Effect of Dry Needling With Electrical Stimulation on Individuals With Restless Legs Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ray M. Lunasin, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-009645
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling with electrical stimulation (Experimental): Participants with restless legs syndrome will receive dry needling with electrical stimulation to the lower extremities
  Interventions: Procedure: Dry Needling with electrical stimulation

INTERVENTIONS:
Procedure: Dry Needling with electrical stimulation — Administered for a total of 2 sessions at a frequency of once per week. The target muscles to be needled will include the gastronemius, soleus, vastus lateralis, rectus femoris, anterior tibialis, posterior tibialis, biceps femoris, and gluteus medius.

SUMMARY:
The purpose of this study is to examine the effects of dry needling with electrical stimulation (DNES) on sleep quality, symptom severity, and function in individuals with restless legs syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Clinical diagnosis of restless legs syndrome

Exclusion Criteria:

* Active cancer diagnoses
* Neuropathic pain (e.g., lumbosacral radiculopathy and/or diabetic neuropathy),
* Pregnancy
* Immunocompromised disease (e.g., HIV, AIDS, lupus)
* Insufficient English-language skills to complete all questionnaires
* Inability to maintain treatment positions
* Contraindications to dry needling:35,36

  * Presence of needle phobia
  * History of abnormal reaction to needling or injection
  * History of bleeding disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality | Baseline, 4 weeks and 8 weeks post-intervention
  Measured using the Pittsburgh Sleep Quality Index (PSQI). Self-report questionnaire that measures general sleep quality. The scoring range is 0-21 with 0-3 scoring for each component. Higher scores indicate worse sleep quality.
Change in periodic limb movement | Baseline, weekly for 3 weeks
  Measured using a consumer-grade sleep tracking device.
Change in Restless Legs Syndrome symptom severity | Baseline, 4 weeks and 8 weeks post-intervention
  RLS symptom severity of each participant will be indexed with likert scale ratings and subacutely by completion of the International Restless Legs Syndrome Rating Scale (IRLSRS). The IRLSRS has demonstrated to be a valid and reliable outcome measure for RLS symptom severity. The scale consists of 10 questions concerning each patient's symptoms and the impact of those symptoms on daily activities and mood. Each question contains answers that score from 0 to 4 points, with 0 representing the absence of a problem and 4 representing a very severe problem. Total scores can range from 0 to 40 with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in pain level | Baseline, 4 weeks and 8 weeks post-intervention
  Measured using the Numerical Pain Rating Scale (NPRS), an 11-point numeric scale ranging from '0' representing "no pain" to '10' representing "worst pain imaginable."
Change in quality of life | Baseline, 4 weeks and 8 weeks post-intervention
  Quality of life will be measured using the EuroQol (EQ-5D-5L), a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on a scale that describes the degree of problems in that area. This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable. The EuroQol has been identified as a valid and reliable outcome measurement for quality of life.
Acute change in Restless Legs Syndrome symptoms | Baseline, Immediately post-intervention
  Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ray Lunasin, PT, DPT, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No